CLINICAL TRIAL: NCT07293650
Title: PREcision MEDicine In Achalasia - A Multicenter Randomized Non-Inferiority Clinical Trial of Short Tailored POEM vs. Standard POEM for Non-Spastic Achalasia and A Multicenter Prospective Cohort Study of Long Tailored POEM for Spastic Esophageal Motility Disorders
Brief Title: PREcision MEDicine In Achalasia (PREMEDIA)
Acronym: PREMEDIA
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Northwestern University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, John Pandolfino, PRINCIPAL INVESTIGATOR (Contact PI), Northwestern University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PREMEDIA (Pro00083748) - 01
Record Dates: First submitted 2025-12-17; First posted 2025-12-19 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Type I Achalasia; Type II Achalasia; EGJ Outflow Obstruction Without Spastic/Hypercontractile Features
Keywords: achalasia; EGJOO
MeSH Terms: conditions — Esophageal Achalasia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard Myotomy (Active Comparator)
  Interventions: Procedure: Standard Myotomy
- Tailored Short Myotomy (Experimental)
  Interventions: Procedure: Tailored Short Myotomy

INTERVENTIONS:
Procedure: Standard Myotomy — Myotomy during POEM of 8-10 cm in length, extending 2-3 cm into the gastric cardia; intention to perform selective circular myotomy, but allowing full thickness myotomy. FLIP is used to confirm adequate myotomy.
  Arms: Standard Myotomy
Procedure: Tailored Short Myotomy — Myotomy during POEM of 4-5 cm in length, extending 1-2 cm into the gastric cardia; intend to perform selective circular myotomy, but allowing full thickness myotomy. FLIP is used to confirm adequate myotomy.
  Arms: Tailored Short Myotomy

SUMMARY:
The goal of this clinical trial is to learn if shorter Per-Oral Endoscopic Myotomy (POEM) works as well as a longer POEM in patients with trouble swallowing due to certain conditions. The main question[s] it aims to answer [is/are]:

* Does making a smaller cut in the muscle at the bottom of the esophagus work just as well as making the standard bigger cut in relieving symptoms?
* Does making the smaller cut reduce the side effects of the procedure compared to the standard bigger cut? Researchers will compare the symptoms and side effects of making a shorter cut to the symptoms and side effects of a longer cut.

Participants will allow researchers to access their standard of care information in their medical record, complete questionnaires at up to 6 times over a 2-year period.

DETAILED DESCRIPTION:
The investigators will perform a randomized controlled trial to compare two different approaches to Peroral Endoscopic Myotomy (POEM) for treating achalasia (Types I and II) and esophagogastric junction outflow obstruction (EGJOO). The most widely used treatment for achalasia is POEM but the current approach involves a 9 cm (3.5 inch) myotomy (cutting of the muscle) to open up the tight lower esophageal sphincter to promote food delivery from the esophagus to the stomach. This approach is very effective, with success rates of approximately 90% over the short term. However, the investigators believe that POEM does not require a full 9 cm myotomy and that the investigators can cut much less muscle (approximately 4cm/1.25inches) to achieve similar improvement in symptoms but with less long-term complications. Cutting less muscle may result in less acid reflux, which is the Achilles heel of any successful treatment for achalasia. A shorter muscle cut may also result in less of a complication known as blown-out myotomy, which causes failure of the esophagus to empty its contents and is a major cause of long-term symptom relapse. The investigators have designed this study to determine whether the shorter myotomy (4 cm) is equivalent to the longer myotomy (9 cm) in terms if symptom improvement, but with the possibility of less acid reflux and blown-out myotomy.

Given these questions, the investigators will enroll 370 patients in a randomized trial where patients will receive either the short tailored (4cm/1.25 inches) or the standard myotomy (9cm/3.5 inches). All patients will undergo intraoperative assessment of success of the myotomy by using a special tool called the functional lumen imaging probe (FLIP). The FLIP will measure the opening dimensions of the lower esophageal sphincter and ensure that the myotomy is adequately performed so that the lower esophageal sphincter can open to a level that will improve esophageal emptying/swallowing. The investigators will follow patients for 2 years in a manner similar to how the investigators would follow patients after achalasia treatment in standard clinical practice. The investigators will assess whether symptoms are similar and whether or not there are differences in acid reflux and esophageal emptying. Patients will undergo follow up testing with questionnaires at intervals of 3-6 months over two years and they will have reflux testing (measure acid exposure using a capsule placed during endoscopy) between 6-12 months and a barium esophagram (X ray while drinking barium) at 2 years. The most important aim is to prove that the symptoms and outcomes success/failure) between the two approaches are similar (short myotomy is non-inferior) and the Eckardt score will be the primary questionnaire score for this study. The investigators believe that this study will help define the optimal approach to POEM in achalasia and also help us prevent complications in the future.

Additionally, the investigators will also ask participants to provide a sample of the muscle tissue that is typically cut during the POEM. This tissue will help us develop a tissue bank to help other researchers looking into the causes of why achalasia and these other esophageal diseases occur. The participants can opt out of this part and still continue in the randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria

1. Age ≥ 18
2. Type I achalasia or type II achalasia or cEGJOO
3. Eckardt score > 3

Exclusion Criteria

The following exclusion criteria are for the RCT, but 1-13 below also pertain to the observational study:

1. Prior POEM
2. Prior surgical treatment for achalasia
3. Endoscopic pneumatic dilation or lower esophageal sphincter botulinum toxin (botox) injection within 6 months
4. Prior unrelated esophageal or upper gastric surgery, including Roux-en-Y gastric bypass and sleeve gastrectomy
5. Prior endoscopic gastroesophageal intervention for obesity or GERD, such endoscopic sleeve gastroplasty or transoral incisionless fundoplication
6. Known secondary achalasia related to malignancy (pseudoachalasia)
7. Known eosinophilic esophagitis
8. Diverticulum (> 2 cm) in distal esophagus
9. Megaesophagus
10. Fibroinflammatory stricture of the esophagus due to any etiology (e.g., peptic, radiation, eosinophilic)
11. Pregnancy
12. Standard contraindications to general anesthesia
13. Standard contraindications to endoscopic myotomy in the esophagus (e.g. untreated varices)
14. Unwillingness or inability to consent for the study
15. Anticipated inability to follow protocol
16. Weekly (or more frequent) opioid medication use in the last 2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 372 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2029-04-01 (Estimated); Study Completion 2030-03-01 (Estimated)

PRIMARY OUTCOMES:
Clinical Response-Overall | From enrollment to Year 2
  Clinical Response is defined by the Eckardt score (a 4-item self-report scale measuring weight loss, chest pain, regurgitation, and dysphagia) with no need for retreatment in 2 years.
Clinical Response-by Sex | From enrollment to Year 2
  Clinical Response is defined by the Eckardt score (a 4-item self-report scale measuring weight loss, chest pain, regurgitation, and dysphagia) with no need for retreatment in 2 years.
Clinical Response-by Race | From Enrollment to Year 2
  Clinical Response is defined by the Eckardt score (a 4-item self-report scale measuring weight loss, chest pain, regurgitation, and dysphagia) with no need for retreatment in 2 years.
Clinical Response-by Ethnicity | From Enrollment to Year 2
  Clinical Response is defined by the Eckardt score (a 4-item self-report scale measuring weight loss, chest pain, regurgitation, and dysphagia) with no need for retreatment in 2 years.

CONTACTS AND LOCATIONS:
Locations (13):
- United States (13):
  - Mayo Clinic Arizona, Scottsdale, Arizona
  - University of California San Diego, La Jolla, California
  - University of Colorado Denver, Denver, Colorado
  - University of Florida, Gainesville, Florida
  - Adventist Health System/Sunbelt, Inc, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - Northwestern University, Chicago, Illinois
  - Johns Hopkins University, Baltimore, Maryland
  - Washington University, St Louis, Missouri
  - Weill Cornell Medical College, New York, New York
  - Case Western Reserve University, Cleveland, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Scott & White Health, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR